CLINICAL TRIAL: NCT05864313
Title: Gaze and Gait Training With Neuromodulation
Brief Title: Gaze and Gait Training With rTMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB202300184
Record Dates: First submitted 2023-03-20; First posted 2023-05-18 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Real 10 Hz rTMS (Active Comparator): Participants will receive 1 hour of real rTMS followed by 1 hour of gaze and gait training.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Gait training; Behavioral: Gaze training
- sham rTMS (Sham Comparator): Participants will receive 1 hour of sham rTMS followed by 1 hour of gaze and gait training.
  Interventions: Behavioral: Gait training; Behavioral: Gaze training; Device: Sham rTMS

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — 10 Hz rTMS for 5 seconds over the frontal eye fields with 25 second intertrain interval for 10 trains (500 pulses) at 90% of the resting motor threshold,
  Other Names: 10 Hz rTMS FEF
  Arms: Real 10 Hz rTMS
Behavioral: Gait training — Subjects will practice stepping on virtual targets with real-time feedback of their foot position displayed on a screen while walking on a treadmill.
Behavioral: Gaze training — Subjects will perform gaze stabilization and gaze shifting exercise via a virtual reality headset.
Device: Sham rTMS — Sham rTMS stimulation will produce discharge noise and vibration without stimulating the cerebral cortex.
  Arms: sham rTMS

SUMMARY:
The purpose of this study is to evaluate the feasibility of combining repetitive transcranial magnetic stimulation (rTMS), gaze and gait training to improve walking and balance in people with or without mild cognitive impairment.

DETAILED DESCRIPTION:
The study plan is to recruit a total of 15 cognitively impaired and 15 healthy adults. The study will involve two visits. Each study visit will involve:

* Real rTMS or sham rTMS that last about 60 minutes
* Gaze stabilization exercise via a virtual reality headset for about 1-hour
* Target stepping on a treadmill for about 1-hour

Researchers will compare changes in gaze and gait following training sessions with real rTMS and sham rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years
* Capable of providing informed consent and complying to the experimental procedures

Exclusion Criteria:

* Significant gait difficulty requiring ambulatory aids
* Presence of implanted device such as a neurostimulator, cochlear implant or pacemaker
* History of epilepsy
* History of hearing issues

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in Foot Placement Error from baseline 1 | Beginning and end of Visit 1, an average of 8 hours
  Foot position relative to stepping targets.
Change in VOR Gain from baseline 1 | Beginning and end of Visit 1, an average of 8 hours
  The amount of eye relative to head movement during active head rotations.
Change in Foot Placement Error from baseline 2 | Beginning and end of Visit 2, an average of 8 hours
  Foot position relative to stepping targets.
Change in VOR Gain from baseline 2 | Beginning and end of Visit 2, an average of 8 hours
  The amount of eye relative to head movement during active head rotations.

SECONDARY OUTCOMES:
Change in Timed Up and Go (TUG) from baseline 1 | Beginning and end of Visit 1, an average of 8 hours
  The TUG assesses mobility, balance, waking ability and fall risk in older adults.
  A higher risk for falling is indicated by >= 12 seconds to complete the test.
Change in Timed Up and Go (TUG) from baseline 2 | Beginning and end of Visit 2, an average of 8 hours
  The TUG assesses mobility, balance, waking ability and fall risk in older adults.
  A higher risk for falling is indicated by >= 12 seconds to complete the test.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Choi, Ph.D., Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No